CLINICAL TRIAL: NCT03586154
Title: Combined Platelet Rich Plasma Intra-articular Shoulder Injection and Stellate Ganglion Block. A New Technique for Management of Chronic Post-mastectomy Shoulder Pain Syndrome
Brief Title: Combined Intra-articular Shoulder Injection and Stellate Ganglion Block in Chronic Post-mastectomy Shoulder Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, Principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MansouraU Nevert
Record Dates: First submitted 2018-06-29; First posted 2018-07-13 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Breast Neoplasms
Keywords: Ketamine; pain; platelet rich plasma; mastectomy; shoulder
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Ketamine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigators were not allowed to know randomization codes and block size until all calculations and measurements had been entered into the database for all patients. All medical caregivers, investigators and patients were blinded to group allocation. One hour before the injection procedure of an enrolled patient, a nurse (not otherwise participating in the study) opened a sealed opaque envelope containing group allocation, and then filled the assigned drug injection for each patient according to the protocol of randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): patients were subjected to ultrasound guided SGB using 1 ml ketamine in a dose of 0.5mg/kg plus 5ml bupivacaine 0.5% in total volume 10 ml
  Interventions: Drug: ketamine and bupivacaine injection
- Group B (Active Comparator): patients were subjected to ultrasound guided SGB using 1 ml ketamine in a dose of 0.5mg/kg plus 5ml bupivacaine 0.5% in total volume 10 ml plus posterior approach shoulder injection with PRP.
  Interventions: Combination Product: Platelet rich plasma; Drug: ketamine and bupivacaine injection

INTERVENTIONS:
Combination Product: Platelet rich plasma — combined platelet rich plasma and 1 ml ketamine in a dose of o.5 ml/kg plus 5ml bupivacaine 0.5% in a total volume 10 ml
  Other Names: PRP
  Arms: Group B
Drug: ketamine and bupivacaine injection — 1 ml ketamine in a dose of o.5 ml/kg plus 5ml bupivacaine 0.5% in a total volume 10 ml

SUMMARY:
Background and Purpose: Adhesive capsulitis of the shoulder is commonly found in patients after breast cancer treatment. We aimed to determine the effectiveness of combined shoulder joint intra-articular injection of platelet rich plasma (PRP) with stellate ganglion block (SGB) with ketamine &bupivacaine injection as a new technique for frozen shoulder (FS) management after mastectomy.

Methods: Sixty four patients with chronic post-mastectomy shoulder pain and stiffness were randomly allocated into one of two groups: group A; ultrasound guided SGB (1 ml ketamine in a dose of 0.5mg/kg plus 5ml bupivacaine 0.5% in total volume 10 ml) and group B; ultrasound guided SGB plus posterior approach shoulder injection with PRP. Visual analogue score (VAS) at rest and at shoulder movement, range of motions (ROM) of shoulder and disability of arm, shoulder and hand (DASH) questionnaire were recorded.

DETAILED DESCRIPTION:
Introduction:

Pain after breast surgery is a significant complication and can persist for several months up to years.The most common sites for pain localization are the axilla, medial upper arm and or lateral / anterior chest wall. Pain can be severe enough to cause long-term disabilities leading to shoulder adhesive capsulitis (frozen shoulder) or complex regional pain syndrome. Of course, this could also interfere with daily activities and sleep leading to negative influence on the quality of life of the affected women. Scar formation, protective posture and tension of the soft tissue after surgery can also cause alteration of the shoulder girdle alignment and immobility.

Adhesive capsulitis of the shoulder is commonly found in breast cancer patients with a prevalence can be as high as 86%.Adhesive capsulitis of the shoulder joint is one of the main producers of Post-mastectomy chronic shoulder pain syndrome , the shoulder joint becomes tight due to capsular inflammation resulting in painful and global ROM restriction. Frozen shoulder management has focused around prolonged courses of physiotherapy to maintain shoulder mobility. Corticosteroids and anti-inflammatory medications are also considered as adjuvant therapies in reducing pain and inflammation.

The stellate ganglion is a nerve bundle related to the sympathetic nervous system providing sensation to the upper body. It is present on either side of the trachea at the 7th cervical vertebrae. The stellate ganglion has second and third order neurons that modulate neuropathic pain to the central nervous system and body temperature. The stellate ganglion block (SGB) is mainly indicated for management of chronic neuropathic painful disorders of the head and neck, upper limb, and upper chest by reducing levels of nerve growth factor leading to a decrease in norepinephrine level that plays a fundamental role in pain transmission in these cases. Ketamine enhances the effect of sympathetic blockade with relief of pain, ischaemia and maintains circulation. And so, ketamine is a useful adjuvant to STGB and it clarify the need of permanent destruction of the ganglion by chemical/ radiofrequency neurolysis in patients with peripheral vascular disease.

Recently, platelet-rich plasma (PRP) have been used in treatment of many soft tissue disorders with positive results being rich in several growth factors and other cytokines that can stimulate healing of soft tissues and joints.

In current study, we aimed to clarify the effectiveness of combined intra-articular PRP injection in shoulder joint with SGB over SGB alone in the challenge of management of post-mastectomy chronic shoulder pain.

Patients and methods:

Study design and participants Our study was a randomized controlled double-blind trial conducted in Anesthesia Department of Medical Faculty and Pain Clinics of Mansoura Oncology Center, Egypt during the period from August 2017 till April 2018. The study was accepted by Institutional Research Board of Mansoura University (Code No: R∕ 17.08.44) and followed the 2008 Helsinki declaration ethical standards.

Seventy patients were assessed for eligibility. Six patients were excluded from the study (four did not meet the inclusion criteria and two declined to participate in the study) (Figure 1). Sixty four patients were included with age of 18 to less than 65 ys who showed post-mastectomy shoulder pain.

Exclusion criteria were patient refusal to participate, Patients with acute shoulder pain (trauma, acute postsurgical pain), secondary adhesive capsulitis (prior surgery or non-surgically induced states of shoulder affection by adhesive capsulitis), hypersensitivity to amide local anesthetics, general contraindications to SGB and cardiac and hepatic, renal or respiratory failure. Written informed consents were obtained from individual participants included in the study.

Sample size It was assessed using G-power analysis. Assuming α (type I error) = 0.05 and β (type II error) = 0.2 (power = 80 %) yielded a total sample size of 70.

Randomization Each patient was assigned in a double-blinded manner to one of two groups. Group A (n=32) patients were subjected to ultrasound guided SGB using 1 ml ketamine in a dose of 0.5mg/kg plus 5ml bupivacaine 0.5% in total volume 10 ml.[9] While group B (n=32) patients were subjected to ultrasound guided SGB using ketamine and bupivacaine in the same dose as group A plus posterior approach shoulder injection with PRP.

An individual not involved in the patient care or data collection randomly assigned the patients using Research Randomizer program into two blocks; each of block size 32 was also randomized using two lists of random numbers. Investigators were not allowed to know randomization codes and block size until all calculations and measurements had been entered into the database for all patients. All medical caregivers, investigators and patients were blinded to group allocation. One hour before the injection procedure of an enrolled patient, a nurse (not otherwise participating in the study) opened a sealed opaque envelope containing group allocation, and then filled the assigned drug injection for each patient according to the protocol of randomization. All data were entered in the database before entering the codes of randomization. The principles for intention-to-treat analysis were followed.

Level of evidence:

Level IV, clinical study

Technique Management and Equipment:

All suitable resuscitation drugs (eg. atropine and adrenaline) and equipment's were available including lipid emulsion for local anesthetic toxicity, endotracheal tubes of different sizes, ambo bag, and ventilator. Under strict aseptic technique for place, patients, and instruments, the different blocks technique done in the operative theater with IV access in place, O2 Mask 6L/minute, and full basic monitoring (Noninvasive Blood Pressure Amplifier, pulse oximeter, and ECG) attached, then all patients in this study were monitored throughout the procedure and up to one hour after the block performance.

Stellate ganglion block technique The anterior para-tracheal approach C6 was done. The patient's neck was extended using a pillow under the shoulder while lying in a supine position aiming to keep the esophagus and the transverse process away from each other. Also the patient was asked to open mouth slightly to make the neck muscles more relaxed. Under complete aseptic technique, a linear probe (5-10 MHz) of Siemens Acuson P300 ultrasound machine was initially placed at the cricoid cartilage level. The location of C6 transverse process was determined by the prominent anterior tubercle (Chassaignac's tubercle). Placement of the ultrasound transducer helped to retract the sternocleidomastoid muscle and carotid sheath laterally and the pressure applied by the transducer reduced the distance between the tubercle and skin and to depress the lung dome to avoid occurrence of pneumothorax. A typical sonographic appearance at the C6 level included the anterior tubercle and transverse process of C6, longus capitis muscle, longus colli muscle (LC), carotid artery, and thyroid gland. We inserted a 22-gauge needle and directed towards to the Chassaignac's tubercle then redirected infero-medially towards the body of C6 until reach out of LC muscle while still staying within the prevertebral fascia (figure 2). After negative aspiration for blood and cerebrospinal fluid, ultrasound guided injection of 1 ml ketamine in a dose of 0.5mg/kg plus 5ml bupivacaine 0.5% in total volume 10 ml 10ml volume was used before in a previous study, and was injected in divided doses (injectate volume of 10 ml used to ensure full ganglion blocked and effective spread of the anesthetic agents at the area of the lower cervical sympathetic chain) (figure 3). The solution was allowed to pass caudally toward the stellate ganglion by raising the head of the patient's bed. We confirmed the success of block by the development of Horner's syndrome at side of injection which included ptosis, myosis, facial anhydrosis, enophthalmos and nasal congestion.

Regulations for PRP Preparation:

At the time of treatment, PRP was obtained from a sample of patient's blood. Thirty ml venous blood was drawn to yield 3-5 cc of PRP. Citrate dextrose A (an anticoagulant) was added to prevent platelet activation prior to its use. Preparation of PRP was done by double centrifugation process; an initial centrifugation to separate red blood cells followed by a second centrifugation to concentrate platelets. The whole blood was initially collected in tubes containing anticoagulants. At the initial centrifugation step, whole blood separates into three layers: an upper layer that contains white blood cells and platelets, an intermediate thin layer (buffy coat layer) that is rich in white blood cells, and a bottom layer that consists mostly of red blood cells. For PRP production, both superficial buffy coat and upper layers were transferred to an empty sterile tube. Then the second centrifugation step was done and should be adequate to help in soft pellets formation (erythrocyte platelets) at the bottom of the tube. We removed the upper portion of the volume (platelet-poor plasma). Pellets were homogenized in lower third (5 ml of plasma) to produce PRP.

Posterior approach shoulder injection techniques:

The patient was placed in either the lateral decubitus or sitting position with the ipsilateral hand placed on the contralateral shoulder. The ultrasound probe (frequency 6-13 MHz) was placed just caudal to the acromion over the infraspinatus tendon. The important anatomical points to identify were humeral head, infraspinatus tendon, labrum, and joint capsule. The posterior approach target was between the cartilage of humeral head underneath the capsule and the free edge of labrum. Once the target was obtained, we inserted a 22 gauge needle from lateral to medial direction with in-plane technique (figure 3) then injected PRP.

The two groups were asked to do some stretching exercises at home as finger walk, cross body reach and outward and inward rotations. The patients were explained how to do these exercises and warm up the shoulder before performing the exercises by moist heating pad for 10-15 minutes.

Outcome Variables Primary outcome: Visual analogue score (VAS) was done at rest and at shoulder movement before injection, one, two and three months after injection. VAS was explained to the patients during assessment as 0 equal no pain and 10 equal worst imaginable pain. Shoulder mobility was assessed while the patient was sitting using goniometry. Secondary outcome: 1-ROM was measured in degrees in five position (extension, flexion, and abduction, internal and external rotation) before and one month after injection. 2-Disability of arm, shoulder and hand (DASH) questionnaire was done before injection, one, two and three months after injection.

Statistical analysis:

The collected data were analyzed using Statistical Package of Social Science (SPSS) program for windows (version 16) and Medcalc program. Quantitative parametric data were presented in means and standard deviations (SD) while non-parametric data were presented in median and range. On testing significance of parametric quantitative data, t-test and ANOVA test were used where the later followed by post hoc test. On testing significance of non-parametric data, Mann-Whitny test, Wilcoxon rank test and Kruskal-Wallis test were used where the later followed by post hoc test. Statistically significant results were considered if p value < 0.05. If p values < 0.001, results were considered highly statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* post-mastectomy shoulder pain
* age of 18 to less than 65 years

Exclusion Criteria:

* refusal to participate
* Patients with acute shoulder pain (trauma, acute postsurgical pain)
* secondary adhesive capsulitis (prior surgery or non-surgically induced states of shoulder affection by adhesive capsulitis)
* hypersensitivity to amide local anesthetics
* general contraindications to SGB and cardiac and hepatic, renal or respiratory failure.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Visual analogue score | Before injection and 1, 2, 3 months after injection
  Visual analogue score (VAS) was done at rest and at shoulder movement before injection, one, two and three months after injection. VAS was explained to the patients during assessment as 0 equal no pain and 10 equal worst imaginable pain. Shoulder mobility was assessed while the patient was sitting using goniometry.

SECONDARY OUTCOMES:
Range of motion | Before injection and one month after injection
  It was measured in degrees in five position (extension, flexion, and abduction, internal and external rotation) before and one month after injection.
Disability of arm | Before injection and 1, 2 , 3 months after injection
  shoulder and hand (DASH) questionnaire was done before injection, one, two and three months after injection.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Tahan, MD, Principal Investigator — Professor of Anesthesia, Medical Faculty, Mansoura University
Locations (1):
- MansouraU, Al Mansurah, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macdonald L, Bruce J, Scott NW, Smith WC, Chambers WA. Long-term follow-up of breast cancer survivors with post-mastectomy pain syndrome. Br J Cancer. 2005 Jan 31;92(2):225-30. doi: 10.1038/sj.bjc.6602304. PMID 15655557
- [Background] Waltho D, Rockwell G. Post-breast surgery pain syndrome: establishing a consensus for the definition of post-mastectomy pain syndrome to provide a standardized clinical and research approach - a review of the literature and discussion. Can J Surg. 2016 Sep;59(5):342-50. doi: 10.1503/cjs.000716. PMID 27668333
- [Background] Ebaugh D, Spinelli B, Schmitz KH. Shoulder impairments and their association with symptomatic rotator cuff disease in breast cancer survivors. Med Hypotheses. 2011 Oct;77(4):481-7. doi: 10.1016/j.mehy.2011.06.015. Epub 2011 Jul 18. PMID 21764521
- [Background] Leonidou A, Woods DA. A preliminary study of manipulation under anaesthesia for secondary frozen shoulder following breast cancer treatment. Ann R Coll Surg Engl. 2014 Mar;96(2):111-5. doi: 10.1308/003588414X13824511649652. PMID 24780667
- [Background] Yang S, Park DH, Ahn SH, Kim J, Lee JW, Han JY, Kim DK, Jeon JY, Choi KH, Kim W. Prevalence and risk factors of adhesive capsulitis of the shoulder after breast cancer treatment. Support Care Cancer. 2017 Apr;25(4):1317-1322. doi: 10.1007/s00520-016-3532-4. Epub 2016 Dec 9. PMID 27942856
- [Background] Aslani H, Nourbakhsh ST, Zafarani Z, Ahmadi-Bani M, Ananloo ME, Beigy M, Salehi S. Platelet-Rich Plasma for Frozen Shoulder: A Case Report. Arch Bone Jt Surg. 2016 Jan;4(1):90-3. PMID 26894228
- [Background] Lipov EG, Joshi JR, Sanders S, Slavin KV. A unifying theory linking the prolonged efficacy of the stellate ganglion block for the treatment of chronic regional pain syndrome (CRPS), hot flashes, and posttraumatic stress disorder (PTSD). Med Hypotheses. 2009 Jun;72(6):657-61. doi: 10.1016/j.mehy.2009.01.009. Epub 2009 Feb 23. PMID 19237252
- [Background] Smith PA. Intra-articular Autologous Conditioned Plasma Injections Provide Safe and Efficacious Treatment for Knee Osteoarthritis: An FDA-Sanctioned, Randomized, Double-blind, Placebo-controlled Clinical Trial. Am J Sports Med. 2016 Apr;44(4):884-91. doi: 10.1177/0363546515624678. Epub 2016 Feb 1. PMID 26831629
- [Background] Peng PW, Cheng P. Ultrasound-guided interventional procedures in pain medicine: a review of anatomy, sonoanatomy, and procedures. Part III: shoulder. Reg Anesth Pain Med. 2011 Nov-Dec;36(6):592-605. doi: 10.1097/AAP.0b013e318231e068. PMID 22005657
- [Background] Stubblefield MD, Custodio CM. Upper-extremity pain disorders in breast cancer. Arch Phys Med Rehabil. 2006 Mar;87(3 Suppl 1):S96-9; quiz S100-1. doi: 10.1016/j.apmr.2005.12.017. PMID 16500198
- [Background] Kulkarni KR, Kadam AI, Namazi IJ. Efficacy of stellate ganglion block with an adjuvant ketamine for peripheral vascular disease of the upper limbs. Indian J Anaesth. 2010 Nov;54(6):546-51. doi: 10.4103/0019-5049.72645. PMID 21224973
- See also: Urbaniak GC, Plous S. Research randomizer. Retrieved July. 1997;7:2008. — http://www.randomizer.org/
- See also: Sweeny J, Grossman BJ. Blood collection, storage and component preparation methods. Tech Manual 14th ed Bethesda MD Am Assoc Blood Banks. 2002;955-8. — https://scholar.google.com.eg/scholar?hl=ar&as_sdt=0%2C5&q=Sweeny+J%2C+Grossman+BJ.+Blood+collection%2C+storage+and+component+preparation+methods.+Tech+Manual+14th+ed+Bethesda+MD+Am+Assoc+Blood+Banks.+2002%3B955%E2%80%938.+&btnG=
- See also: Welsh WJ. Autologous platelet gel: clinical function and usage in plastic surgery. Cosmet Derm. 2000;11:13. — https://scholar.google.com.eg/scholar?hl=ar&as_sdt=0%2C5&q=SWelsh+WJ.+Autologous+platelet+gel%3A+clinical+function+and+usage+in+plastic+surgery.+Cosmet+Derm.+2000%3B11%3A13.+&btnG=